CLINICAL TRIAL: NCT02466243
Title: A Phase 2, Double-blind, Randomized, Placebo-controlled Study to Investigate the Safety, Tolerability, and Efficacy of JBT-101 in Subjects With Dermatomyositis
Brief Title: Safety, Tolerability, and Efficacy of JBT-101 in Subjects With Dermatomyositis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor terminated open-label extension.
Sponsor: Corbus Pharmaceuticals Inc. (Industry)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH); University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: JBT101-DM-001; 116313 (Registry Identifier: Investigation New Drug Application (IND)); R21AR066286 (NIH)
Record Dates: First submitted 2015-06-02; First posted 2015-06-09 (Estimated); Results first posted 2023-01-19 (Actual); Last update posted 2023-01-19 (Actual); Status verified 2022-12

CONDITIONS: Dermatomyositis
Keywords: JBT-101, lenabasum, dermatomyositis
MeSH Terms: conditions — Dermatomyositis | interventions — lenabasum

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- JBT-101 (Experimental): Part A: JBT-101 20 mg capsule once a day on Days 1-28, then 20 mg capsule twice a day on Days 29-84.
  Part B: JBT-101 20 mg twice daily on Days 1 - 365 of the OLE.
  Interventions: Drug: JBT-101
- Placebo (Placebo Comparator): Part A: Placebo capsule once a day on Days 1-28, then placebo capsule twice a day on Days 29-84.
  Part B: Placebo twice daily on Days 1 - 365 of the OLE.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: JBT-101 — Part A: 20 mg once daily on Days 1-28, then 20 mg twice daily on Days 29-84.
  Part B: JBT-101 20 mg twice daily on Days 1 - 365 of the OLE.
  Other Names: lenabasum
  Arms: JBT-101
Drug: Placebo — Part A: Once daily on Days 1-28, then twice daily on Days 29-84.
  Part B: Placebo twice daily on Days 1 - 365 of the OLE.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability and efficacy of JBT-101 in adult subjects with skin-predominant, dermatomyositis (DM) that is refractory to at least 3 months treatment with hydroxychloroquine.

DETAILED DESCRIPTION:
Part A: An interventional, double-blind, randomized, placebo-control design will be used to test JBT-101 in about 22 eligible male or female subjects ≥ 18 and ≤ 70 years of age with moderate-to-severe active skin-predominant dermatomyositis.

Part B: A one-year open-label design to test JBT-101 in subjects who completed Part A without permanent discontinuation of study product because of safety or tolerability reasons.

ELIGIBILITY:
Inclusion Criteria (Part A):

* CDASI activity score ≥ 14;
* No difficulty with lifting or walking, and no more than 1.5 x the upper limit of normal of creatine phosphokinase or aldolase;
* Failed at least 3 months treatment with hydroxychloroquine;
* Stable treatment for dermatomyositis for at least 28 days before Visit 1 (Day 1).

Inclusion Criteria (Part B):

* Completion of dosing in Part A without permanent discontinuation of study product because of safety or tolerability reasons

Exclusion Criteria (Part A and B):

* Significant diseases or conditions other than DM that may influence response to the study product or safety;
* Any one of the following values for laboratory tests at Screening:

  1. A positive pregnancy test (or at Visit 1);
  2. Hemoglobin < 10 g/dL;
  3. Neutrophils < 1.0 x 10^9/L;
  4. Platelets < 75 x 10^9/L;
  5. Creatinine clearance < 50 ml/min according to modified Cockcroft-Gault equation;
  6. Aspartate aminotransferase, alanine aminotransferase, or alkaline phosphatase > 2.5 x upper normal limit;
  7. Total bilirubin ≥ 1.5 x upper limit of normal.
* Any other condition that, in the opinion of the Principal Investigator, is clinically significant and may put the subject at greater safety risk, influence response to study product, or interfere with study assessments.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2015-06; Primary Completion 2017-08 (Actual); Study Completion 2021-01-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Victoria Werth, M.D., Principal Investigator — University of Pennsylvania Perlman School of Medicine
Locations (1):
- University of Pennsylvania Perlman School of Medicine, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Stone CJ, Ahuja G, Lopes Almeida Gomes L, Poroye J, Faden DF, Xie L, Feng R, White B, Werth VP. Long-Term Safety and Efficacy of Lenabasum, a Cannabinoid Receptor Type 2 Agonist, in Patients with Dermatomyositis with Refractory Skin Disease: Follow-Up Data from a 3-Year Open-Label Extension Study. JID Innov. 2024 Sep 5;5(1):100311. doi: 10.1016/j.xjidi.2024.100311. eCollection 2025 Jan. PMID 39403556
- [Derived] Werth VP, Hejazi E, Pena SM, Haber J, Zeidi M, Reddy N, Okawa J, Feng R, Bashir MM, Gebre K, Jadoo AS, Concha JSS, Dgetluck N, Constantine S, White B. Safety and Efficacy of Lenabasum, a Cannabinoid Receptor Type 2 Agonist, in Patients with Dermatomyositis with Refractory Skin Disease: A Randomized Clinical Trial. J Invest Dermatol. 2022 Oct;142(10):2651-2659.e1. doi: 10.1016/j.jid.2022.03.029. Epub 2022 Apr 29. PMID 35490744

RESULTS

PARTICIPANT FLOW:
Groups:
- JBT-101: Part A: JBT-101 20 mg capsule once a day on Days 1-28, then 20 mg capsule twice a day on Days 29-84.
  Part B: JBT-101 20 mg twice daily on Days 1 - 365 of the OLE.
  JBT-101: Part A: 20 mg once daily on Days 1-28, then 20 mg twice daily on Days 29-84.
  Part B: JBT-101 20 mg twice daily on Days 1 - 365 of the OLE.
- Placebo: Part A: Placebo capsule once a day on Days 1-28, then placebo capsule twice a day on Days 29-84.
  Part B: Placebo twice daily on Days 1 - 365 of the OLE.
  Placebo: Part A: Once daily on Days 1-28, then twice daily on Days 29-84.
  Part B: Placebo twice daily on Days 1 - 365 of the OLE.
Period: Part A Treatment Period (Double Blind)
Arm/Group | JBT-101 | Placebo
Started | 11 | 11
Completed | 11 | 11
Not Completed | 0 | 0
Period: Part B Open-label Treatment Period
Arm/Group | JBT-101 | Placebo
Started | 11 | 10 (Participant decided not to participate in Part B)
Completed | 0 | 0
Not Completed | 11 | 10
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Sponsor Decision | 8 | 6
Not completed — Missing | 2 | 2

BASELINE CHARACTERISTICS:
Population: Numbers reflect all randomized subjects; all subjects were included in the safety, modified intent-to-treat, and per protocol populations
Groups:
- Total: Total of all reporting groups
Arm/Group | JBT-101 | Placebo | Total
Number analyzed (Participants) | 11 | 11 | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.1 (9.31) | 52.5 (10.44) | 52.8 (9.66)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 11 | 21
  Male | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 0 | 3
  Not Hispanic or Latino | 8 | 11 | 19
  Unknown or Not Reported | 0 | 0 | 0
Race [Count of Participants; unit: Participants] — number of participants by race
  Participants
    White | 11 | 10 | 21
    Black or African American | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change in Cutaneous Dermatomyositis Disease Area and Severity Index (CDASI) From Baseline in Part A.
Description: The CDASI is a validated outcome measure that systematically quantifies cutaneous DM disease activity, In the CDASI, DM skin disease activity is scored from 0 to 100 based on the physician's evaluation of erythema, scale, and erosion or ulceration at 15 anatomic locations as well as alopecia, Gottron's sign or papules on the hands, and periungual changes. A 5-point or greater decrease in the CDASI activity score indicates clinically relevant improvement based on statistical analysis using a receiver operating characteristic curve to maximize sensitivity and specificity
Time Frame: Part A: 84-day treatment period (Change from the Baseline CDSAI score at Day 84)
Population: modified intent-to-treat population LS mean (SE) at Day 84
Measure: Least Squares Mean (Standard Error); unit: CDASI Activity Score
Groups:
- Lenabasum: lenabasum 20 mg BID
- Placebo: Placebo BID
Arm/Group | Lenabasum | Placebo
Number analyzed (Participants) | 11 | 11
CDASI Activity Score | -8.0 (8.16) | -5.5 (5.56)

2. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events as a Measure of Safety and Tolerability
Description: Number of participants with treatment emergent adverse events were assessed as a measure of safety and tolerability
Time Frame: Part A: to Day 84
Population: Safety Population
Measure: Count of Participants; unit: Participants
Groups:
- Lenabasum: Part A: JBT-101 20 mg capsule once a day on Days 1-28, then 20 mg capsule twice a day on Days 29-84.
  JBT-101: Part A: 20 mg once daily on Days 1-28, then 20 mg twice daily on Days 29-84.
- Placebo: Part A: Placebo capsule once a day on Days 1-28, then placebo capsule twice a day on Days 29-84.
  Placebo: Part A: Once daily on Days 1-28, then twice daily on Days 29-84.
Arm/Group | Lenabasum | Placebo
Number analyzed (Participants) | 11 | 11
Participants
  Any TEAE | 11 | 8
  Any serious TEAE | 0 | 0
  Any TEAE leading to discontinuation | 0 | 0
  Any severe TEAE | 0 | 0
  No TEAE | 0 | 3

3. Secondary Outcome: Change in Patient-reported Outcomes From Baseline at 84 Days for Part A
Description: LS mean (SE) change from baseline to Week 6 (Day 84) for lenabasum vs. placebo using a mixed model repeated measures analysis
  The CDASI is a validated outcome measure that systematically quantifies cutaneous DM disease activity and damage, In the CDASI, the Damage Score is scored from 0 to 32 based on the physician's evaluation of poikiloderma and calcinosis. 0 representing no damage and 32 representing the greatest level of damage.
Time Frame: Part A: 84-day treatment period
Population: modified intent to treat population
Measure: Least Squares Mean (Standard Error); unit: CDASI Damage Score
Groups:
- Lenabasum 20 mg BID: Lenabasum 20 mg once daily from Day 1 to Day 28, then 20 mg BID to Day 84
Arm/Group | Placebo | Lenabasum 20 mg BID
Number analyzed (Participants) | 11 | 11
CDASI Damage Score | -5.5 (5.56) | -8.0 (8.16)

ADVERSE EVENTS:
Time Frame: 84 days
Arm/Group | JBT-101 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11
Other Adverse Events (participants affected / at risk) | 11/11 | 11/11
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | JBT-101 (N=11) | Placebo (N=11)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 1 (2)
Dry mouth (Gastrointestinal disorders) | 4 (4) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2)
Fatigue (General disorders) | 1 (1) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 2 (3) | 0 (0)
Increased appetite (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Dizziness (Nervous system disorders) | 5 (8) | 2 (2)
Headache (Nervous system disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-01-03): https://cdn.clinicaltrials.gov/large-docs/43/NCT02466243/Prot_000.pdf
  • Statistical Analysis Plan (2017-09-06): https://cdn.clinicaltrials.gov/large-docs/43/NCT02466243/SAP_001.pdf